CLINICAL TRIAL: NCT03702374
Title: Effect of Prolonged Combined Antioxidant Therapy Intake on Oxidative Stress and Mitochondrial Dysfunction Markers in Patients With Diabetic Retinopathy
Brief Title: Combined Antioxidant Therapy on Oxidative Stress, Mitochondrial Dysfunction Markers in Diabetic Retinopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Adolfo Daniel Rodriguez-Carrizalez, Clinical Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RD-20170102
Record Dates: First submitted 2018-10-02; First posted 2018-10-11 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; oxidative stress; mitochondrial dysfunction; oxidative markers; diabetes; antioxidant therapy
MeSH Terms: conditions — Diabetic Retinopathy; Mitochondrial Diseases; Diabetes Mellitus | interventions — Magnesium Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined Antioxidant Therapy group (Experimental): This arm will be administered with the combined antioxidant therapy, and will consist of 30 patients with moderate non-proliferative diabetic retinopathy (NPDR), 30 subjects with severe NPDR and 30 patients with Proliferative diabetic retinopathy.
  Interventions: Drug: Combined antioxidant therapy
- Placebo group (Placebo Comparator): This arm will be administered with placebo, and will consist of 30 patients with moderate non-proliferative diabetic retinopathy (NPDR), 30 subjects with severe NPDR and 30 patients with Proliferative diabetic retinopathy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Combined antioxidant therapy — It consists in a tablet with lutein (10 mg), astaxanthin (4 mg), Zeaxanthin (1mg), vitamin C (L-ascorbic acid 180mg), vitamin E (DL-alpha tocopherol 30mg), zinc (zinc oxide 20mg), copper (copper sulfate 1mg), taken once a day for 12 months
  Other Names: Drusen Laz
  Arms: Combined Antioxidant Therapy group
Other: Placebo — It consists in a capsule with 100mg of magnesium oxide.
  Other Names: Magnesia
  Arms: Placebo group

SUMMARY:
The present study aims to support previous research on antioxidant therapy effects in diabetic retinopathy outcome. The investigators intend to assess 180 patients with diabetic retinopathy in different stages (moderate, severe and proliferative), whom either will be assigned to placebo group or combined antioxidant therapy. Each group will receive the intervention for 12 months. Such intervention consists in taking one tablet (placebo or antioxidant therapy) orally, a day.

At baseline, blood and urine samples will be collected in order to assess metabolic and oxidative stress status, mitochondrial function or dysfunction, liver and kidney function. In addition, fluorescein angiography will be done for the categorization of diabetic retinopathy. After six months and at the end of the intervention, blood and urine measurements as well as angiographies will be done for comparing the outcomes between both groups and correlate oxidative stress status, mitochondrial dysfunction with grade of retinopathy.

DETAILED DESCRIPTION:
Diabetic retinopathy is a diabetes microvascular complication due to an insufficient oxygen supply to its endothelial cells in states of constant hyperglycemia. This entity is classified in two main categories: non-proliferative diabetic retinopathy and proliferative diabetic retinopathy, the latter is characterized for the presence of neovascularization as oppose to the first one.

Oxidative stress has been considered as one of the main factors in the development of diabetic retinopathy. It results from an imbalance between oxidants production and cellular antioxidant defenses, which provokes DNA damage in the mitochondrion altering its capacity to produce ATP (Adenosine Triphosphate) resulting in what is known as mitochondrial dysfunction.

Diabetic retinopathy management merely comprises glycemic, lipemic and blood pressure control. Secondary intervention includes anti-platelet agents, protein-kinase C inhibitors, aldolase reductase inhibitors, laser and vitrectomy. Antioxidant therapy has been used as a co-adjuvant for these interventions, as antioxidant substances that complement action and efficacy of the established treatment for diabetic retinopathy.

Diabetic retinopathy is the principal cause of blindness in persons between 20 and 70 years of age. Its prevalence is, approximately, 25% 5 years after diagnosis.

Which is why the investigators intend to prove if the antioxidant therapy is able to change retinopathy outcomes in oxidative stress, mitochondrial dysfunction and/or grade of retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes with moderate or severe non-proliferative diabetic retinopathy without clinically significant macular edema.
* Patients with type 2 diabetes with proliferative diabetic retinopathy without clinically significant macular edema.
* In current treatment that may include: metformin, glibenclamide, pravastatin, bezafibrate, losartan, nifedipine or captopril.
* HbA1c equal or lower than 9%
* LDL under 190mg/dl, triglycerides under 500mg/dl)
* Blood pressure under 180/110 mmHg
* Non-smoker or inactive for at least 6 months
* Signed informed consent

Exclusion Criteria:

* Antioxidant therapy intake over the last 6 months. Antioxidant dietary intake that surpasses the daily DIR (dietary intake recommendations)
* Patients who require secondary intervention (laser surgery)
* Patients with previous history of myocardial infarction, ictus or severe peripheral vasculopathy
* Patients with pathologies that increase oxidative stress
* Patients with neurodegenerative or carcinogen processes
* Hepatic or renal failure
* Pregnancy
* Patients with hypersensitivity to therapy components
* Other ocular pathologies, such as cataract, glaucoma, corneal dystrophy, macular degeneration among others
* Patients who are currently participating in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in concentration of serum malondialdehyde after intervention. | 3 measures will be made, 1 at baseline, another one after 6 months and a last one after completion of 12 months of intervention.
  The investigators will consider changes presented in plasma concentrations of malondialdehyde from baseline to the end of the intervention. The investigators expect to find a decrease in malondialdehyde concentrations in the supplemented group.
Changes in ATPase activity after intervention from baseline | 3 measures will be made, 1 at baseline, another one after 6 months and a last one after 12 months of intervention
  The investigators will consider changes showed in ATPase activity after the intervention compared to baseline. The investigators expect to find a decrease in ATPase activity in the supplemented group.
Changes in concentration of total antioxidant capacity (TAC) after intervention from baseline. | 3 measures will be made, 1 at baseline, another one after 6 months and a last one after 12 months of intervention
  The investigators will consider changes presented in plasma concentrations of total antioxidant capacity (TAC) from baseline to the end of the intervention. The investigators expect to find TAC augmentation in the supplemented group.

SECONDARY OUTCOMES:
Diabetic retinopathy severity progress at the end of intervention from baseline | 2 measures will be made, 1 at baseline and a second one after 12 months of intervention.
  Change in grade of retinopathy according to the International Clinical Diabetic Retinopathy Disease Severity Scale.
  No apparent retinopathy: No abnormalities. Mild non-proliferative diabetic retinopathy: presence of microaneurysms only. Moderate non-proliferaitve diabetic retinopathy: More than just microaneurysms but less than Severe Non-proliferative diabetic retinopathy.
  Severe non-proliferative diabetic retinopathy: Presence of more than 20 intraretinal hemorrhages in each of 4 quadrants, venous beading in 2 or more quadrants, prominent intraretinal microvascular anormalities in one or more quadrants, no signs of proliferative retinopathy.
  Proliferative diabetic retinopathy: presence of neovascularization, or vitreous/preretinal hemorrhage.
  Note: Progression from a moderate non-proliferative diabetic retinopathy to a severe non-proliferative diabetic retinopathy, and from either of those two to proliferative retinopathy will be considered as a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo D. Rodriguez-Carrizalez, PhD, Study Director — Clinical Investigator at University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics,, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
The results of this study will be published in an open access journal with impact factor according to Journal Citation Reports. Considering the global clinical status of participants before and after of pharmacological intervention.

REFERENCES:
- [Background] Rodriguez-Carrizalez AD, Castellanos-Gonzalez JA, Martinez-Romero EC, Miller-Arrevillaga G, Villa-Hernandez D, Hernandez-Godinez PP, Ortiz GG, Pacheco-Moises FP, Cardona-Munoz EG, Miranda-Diaz AG. Oxidants, antioxidants and mitochondrial function in non-proliferative diabetic retinopathy. J Diabetes. 2014 Mar;6(2):167-75. doi: 10.1111/1753-0407.12076. Epub 2013 Aug 21. PMID 23875878
- [Background] Rodriguez-Carrizalez AD, Castellanos-Gonzalez JA, Martinez-Romero EC, Miller-Arrevillaga G, Roman-Pintos LM, Pacheco-Moises FP, Miranda-Diaz AG. The antioxidant effect of ubiquinone and combined therapy on mitochondrial function in blood cells in non-proliferative diabetic retinopathy: A randomized, double-blind, phase IIa, placebo-controlled study. Redox Rep. 2016 Jul;21(4):190-5. doi: 10.1179/1351000215Y.0000000032. Epub 2016 Feb 5. PMID 26207797
- [Background] Rodriguez-Carrizalez AD, Castellanos-Gonzalez JA, Martinez-Romero EC, Miller-Arrevillaga G, Pacheco-Moises FP, Roman-Pintos LM, Miranda-Diaz AG. The effect of ubiquinone and combined antioxidant therapy on oxidative stress markers in non-proliferative diabetic retinopathy: A phase IIa, randomized, double-blind, and placebo-controlled study. Redox Rep. 2016 Jul;21(4):155-63. doi: 10.1179/1351000215Y.0000000040. Epub 2015 Aug 31. PMID 26321469
- [Background] Sonia Sifuentes-Franco, Adolfo Daniel Rodríguez-Carrizalez, Sandra Carrillo- Ibarra, José Alberto Castellanos-González, Esaú César Martínez-Romero, Guillermo Miller-Arrevillaga and Alejandra Guillermina Miranda-Díaz. The effect of Ubiquinone administration on oxidative DNA damage and repair in plasma levels in non-proliferative diabetic retinopathy.Diabetes Management 2017;7(2):186-191
- [Background] Lopez-Contreras AK, Martinez-Ruiz MG, Olvera-Montano C, Robles-Rivera RR, Arevalo-Simental DE, Castellanos-Gonzalez JA, Hernandez-Chavez A, Huerta-Olvera SG, Cardona-Munoz EG, Rodriguez-Carrizalez AD. Importance of the Use of Oxidative Stress Biomarkers and Inflammatory Profile in Aqueous and Vitreous Humor in Diabetic Retinopathy. Antioxidants (Basel). 2020 Sep 20;9(9):891. doi: 10.3390/antiox9090891. PMID 32962301
- [Background] Robles-Rivera RR, Castellanos-Gonzalez JA, Olvera-Montano C, Flores-Martin RA, Lopez-Contreras AK, Arevalo-Simental DE, Cardona-Munoz EG, Roman-Pintos LM, Rodriguez-Carrizalez AD. Adjuvant Therapies in Diabetic Retinopathy as an Early Approach to Delay Its Progression: The Importance of Oxidative Stress and Inflammation. Oxid Med Cell Longev. 2020 Mar 11;2020:3096470. doi: 10.1155/2020/3096470. eCollection 2020. PMID 32256949
- [Background] Cecilia OM, Jose Alberto CG, Jose NP, Ernesto German CM, Ana Karen LC, Luis Miguel RP, Ricardo Raul RR, Adolfo Daniel RC. Oxidative Stress as the Main Target in Diabetic Retinopathy Pathophysiology. J Diabetes Res. 2019 Aug 14;2019:8562408. doi: 10.1155/2019/8562408. eCollection 2019. PMID 31511825